CLINICAL TRIAL: NCT01046240
Title: Randomized Crossover Pharmacokinetic Evaluation of Subcutaneous (SC) Versus Intravenous Palonosetron in Cancer Patients Treated With Platinum Based Chemotherapy
Brief Title: Pharmacokinetic Evaluation of Subcutaneous Versus Intravenous Palonosetron in Cancer Treated With Chemotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PAL/SC-IV-2008; 2008-002853-19 (EudraCT Number)
Record Dates: First submitted 2009-11-24; First posted 2010-01-11 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2012-11

CONDITIONS: Emesis
Keywords: chemotherapy; emesis; palonosetron
MeSH Terms: conditions — Vomiting | interventions — Palonosetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous palonosetron (Active Comparator): Intravenous palonosetron: control arm (standard treatment)
  Interventions: Drug: Palonosetron
- subcutaneous palonosetron (Experimental): subcutaneous palonosetron
  Interventions: Drug: Palonosetron

INTERVENTIONS:
Drug: Palonosetron — Palonosetron 3 mg administered SC or IV

SUMMARY:
This trial compares the pharmacokinetics of palonosetron administered subcutaneously and intravenously.

DETAILED DESCRIPTION:
5-Hydroxitryptamine3 antagonists are one of the mainstays of antiemetic treatment and they are administered either intravenously or orally. Nevertheless sometimes neither administration route is feasible, such as in patients unable to admit oral intake managed in an outpatient setting. Our objective is to evaluate the bioavailability of subcutaneous palonosetron.Patients receiving platinum-based chemotherapy will be randomized to receive palonosetron 3 mg either subcutaneously or intravenously in a crossover manner during two cycles. Blood and urine samples will be collected after each cycle. Pharmacokinetics of subcutaneous and IV palonosetron will be prospectively compared.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients receiving platinum-based chemotherapy adequate bone marrow, hepatic and renal function

Exclusion Criteria:

* Pregnancy
* Serious concomitant diseases, in the invesgator´s criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To assess the pharmacokinetics of a single dose of palonosetron 3mg administered either subcutaneously or intravenously by assessment of area under the curve and Cmax in cancer patients treated with emetogenic chemotherapy. | Palonosetron levels will be assessed at 10 , 15, 30, 45, 60 min. and 12 and 24 hours following treatment

SECONDARY OUTCOMES:
To compare the efficacy of a single dose of palonosetron 3mg administered either subcutaneously or intravenously by assessment of number of episodes of nausea and vomiting in cancer patients treated with emetogenic chemotherapy. | 1 week (post-chemotherapy)

CONTACTS AND LOCATIONS:
Overall Officials: Belen Sadaba, MD, PhD, Principal Investigator — Clinica Universidad de Navarra
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain

REFERENCES:
- [Derived] Sadaba B, del Barrio A, Campanero MA, Azanza JR, Gomez-Guiu A, Lopez-Picazo JM, Algarra SM, Guillen Grima F, Blanco Prieto M, Perez-Gracia JL, Gurpide A. Randomized pharmacokinetic study comparing subcutaneous and intravenous palonosetron in cancer patients treated with platinum based chemotherapy. PLoS One. 2014 Feb 27;9(2):e89747. doi: 10.1371/journal.pone.0089747. eCollection 2014. PMID 24587006